CLINICAL TRIAL: NCT06207422
Title: The Effects of a Moderate Intensity Training Program Versus a High Intensity Training Program on Central Pain Processing
Acronym: ChronicPA-PAIN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated prematurely due to difficulties in participant recruitment. We reframed the project as a pilot feasibility study to better assess recruitment processes and inform the design of a future full-scale trial.
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ONZ-2023-0425
Record Dates: First submitted 2023-12-18; First posted 2024-01-17 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: moderate intensity training; high intensity training; pressure pain threshold; conditioned pain modulation; exercise induced hypoalgesia; nociceptive flexion reflex; quantitative sensory testing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Moderate intensity training program (Experimental)
  Interventions: Other: Moderate intensity training program
- High intensity training program (Experimental)
  Interventions: Other: High intensity training program

INTERVENTIONS:
Other: Moderate intensity training program — A 10-week intervention program performed at 60-70% of the heart rate reserve. Heart rate reserve will be calculated using the Karvonen formula (target heart rate = [(predicted maximum heart rate (= 220 - age) - resting heart rate) x %intensity] + resting heart rate). The intervention program will consist of three exercise sessions per week, of which one guided group session at Ghent University Hospital and two sessions to be carried out at home.
  Arms: Moderate intensity training program
Other: High intensity training program — A 10-week intervention program performed at ≥80% of the predicted maximum heart rate (target heart rate = predicted maximum heart rate (= 220 - age) x %intensity). The intervention program will consist of three exercise sessions per week, of which one guided group session at Ghent University Hospital and two sessions to be carried out at home.
  Arms: High intensity training program

SUMMARY:
Previous studies have shown that healthy individuals who take more steps per day and who spend more time on moderate- to vigorous-intensity activities exhibit better pain inhibition and less pain facilitation. Furthermore, exercise training (i.e., exercise performed over a number of sessions) can result in reduced pain sensitivity (increased pressure pain threshold). However, the optimal exercise prescription required to achieve pain sensitivity reduction is currently unclear. The next step is to determine experimentally whether increasing physical fitness will lead to positive effects on central pain processing (i.e., pain sensitivity, pain modulation, spinal nociception). The aim of this study is to examine the effects of two exercise programs on central pain processing in healthy sedentary individuals. In case of positive effects, this would provide a rationale for the future to investigate this in chronic pain patients with impaired pain modulation.

DETAILED DESCRIPTION:
Objectives:

Since research on the effects of chronic exercise interventions on pain modulation is scarce and since there is no optimal exercise prescription to reduce pain sensitivity, the effects of a moderate intensity training (MIT) program versus a high intensity training (HIT) program on central pain processing will be examined in healthy sedentary individuals.

Study population:

Thirty healthy sedentary adults between 18 and 55 years of age and with a body mass index (BMI) between 20 and 25 kg/cm² will be recruited. Sedentary is defined as "having a sedentary job and performing less than three hours of moderate physical activity per week". Moderate physical activity is defined as "an activity that requires at least three times the amount of passively expended energy". The sample size was calculated based on a similar previously conducted study.

Study Protocol:

The participants will be invited for a first contact moment (T0) at Ghent University Hospital or at the participant's homes. During T0, participants will be asked to sign an informed consent form. Furthermore, the procedure of the intervention will be explained and a general questionnaire on sociodemographic and health-related characteristics will be administered. Participants will then receive an ActiGraph accelerometer to take home and wear for seven consecutive days to monitor physical activity (i.e., number of steps, moderate and vigorous physical activity, and sedentary behavior).

After wearing the Actigraph accelerometer for seven consecutive days, participants will be invited for a first test moment (T1) at Ghent University Hospital. During T1, three questionnaires will be administered, namely a day survey (intake of medication, caffeine, alcohol and nicotine in the past 24 hours and performance of extreme physical exertion in the past 48 hours), the International Physical Activity Questionnaire (IPAQ) and the Hospital Anxiety and Depression Scale (HADS). Before the start of the experimental pain measurements, blood pressure will be measured with a blood pressure monitor and resting heart rate will be measured using a heart rate belt around the chest.

Next, central pain processing will be assessed:

1. to evaluate pain sensitivity, pressure algometry will be performed using a digital algometer to determine the pressure pain threshold (PPT) bilaterally on the muscle belly of the extensor carpi radialis and the rectus femoris.
2. to evaluate pain inhibition, a conditioned pain modulation (CPM) paradigm will be performed in which the measurement of the PPT (= test stimulus (TS)) will be repeated on the dominant body side during (at minute two) and two minutes after immersion of the non-dominant hand in a warm water bath (= conditioning stimulus (CS)) of 45.5°C for six minutes.
3. to evaluate exercise-induced hypoalgesia (EIH), the PPT measurements will be repeated before (bilaterally) and after (on the dominant body side) a submaximal exercise test (Aerobic Power Index test) performed on an electrically braked bicycle ergometer. Cycling will start at a load of 25 W. Then the load will be increased by 25 W every minute until the submaximal level, defined as 75% of the predicted maximum heart rate (= 220 - age), is reached. Heart rate will be measured before, during, and after the test with a heart rate belt around the chest.
4. to evaluate spinal nociception, transcutaneous electrical neurostimulation (TENS) of the n. suralis of the dominant leg will be performed using a bar electrode. The nociceptive flexion reflex (NFR) threshold will be determined, as well as the pain intensity during repetitive stimulation at the intensity of the NFR threshold to evaluate temporal summation of the NFR. The elicitation of the NFR will be evaluated by measuring the involuntary contraction of the ipsilateral biceps femoris, which will be recorded using electromyography (EMG).

After the experimental pain measurements, the test subjects will receive a Fitbit smartwatch to measure weekly step count during the 10-week exercise program.

After T1, the participants will be randomly assigned to one of two 10-week intervention programs, namely a MIT or a HIT program based on a 1:1 ratio.

Upon completion of the intervention, participants' physical activity will be monitored again for 7 consecutive days using an Actigraph accelerometer. After these 7 days, participants will be invited again for a second test moment (T2) at Ghent University Hospital. During T2, the day survey and the IPAQ will be administered again, blood pressure will be measured and the pain measurements will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 55 years
* BMI between 20 and 25 kg/m²
* Dutch-speaking
* sedentary job and performing less than 3 hours of moderate physical activity per week

Exclusion Criteria:

* current pain complaints or other (medical and/or psychological) health problems
* history of serious pain complaints or (medical and/or psychological) health problems
* history of serious conditions (e.g. cancer, cardiovascular disease, epilepsy, diabetes, depression, etc.)
* being pregnant
* pregnant in the past 12 months
* currently breastfeeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2024-08-23 (Actual)

PRIMARY OUTCOMES:
Pressure pain threshold | Change from baseline (T1) at 1 week after intervention (T2)
  Pressure algometry will be performed using a digital algometer to determine the pressure pain threshold bilaterally on the muscle belly of the extensor carpi radialis and the rectus femoris.
Conditioned pain modulation | Change from baseline (T1) at 1 week after intervention (T2)
  A conditioned pain modulation paradigm will be performed in which the measurement of the pressure pain threshold (= test stimulus) will be repeated on the dominant body side during (at minute two) and two minutes after immersion of the non-dominant hand in a warm water bath (= conditioning stimulus) of 45.5°C for six minutes.
Exercise-induced hypoalgesia | Change from baseline (T1) at 1 week after intervention (T2)
  To evaluate exercise-induced hypoalgesia, the pressure pain threshold measurements will be repeated before (bilaterally) and after (on the dominant body side) a submaximal exercise test (Aerobic Power Index test) performed on an electrically braked bicycle ergometer.
Nociceptive flexion reflex - threshold | Change from baseline (T1) at 1 week after intervention (T2)
  The nociceptive flexion reflex will be elicited by performing transcutaneous electrical nerve stimulation of the sural nerve of the dominant leg in its retromalleolar path using a bar electrode. The elicitation of the NFR will be evaluated by measuring the involuntary contraction of the ipsilateral biceps femoris, which will be recorded using electromyography.
Nociceptive flexion reflex - temporal summation | Change from baseline (T1) at 1 week after intervention (T2)
  Five 1ms rectangular wave pulse train will be administered 3 times at a frequency of 2 Hz at a constant stimulation intensity. This procedure will be repeated 5 times.

SECONDARY OUTCOMES:
Hospital anxiety and depression scale | Baseline (T1)
  Self-report measure assessing anxiety and depression
International physical activity questionnaire | Change from baseline (T1) at 1 week after intervention (T2)
  Self-report measure assessing physical activity during the previous 7 days
Moderate physical activity | Change from baseline (T1) at 1 week after intervention (T2)
  Moderate physical activity will be measured with an ActiGraph accelerometer during 7 consecutive days.
Vigorous physical activity | Change from baseline (T1) at 1 week after intervention (T2)
  Vigorous physical activity will be measured with an ActiGraph accelerometer during 7 consecutive days.
Sedentary behavior | Change from baseline (T1) at 1 week after intervention (T2)
  Sedentary behavior will be measured with an ActiGraph accelerometer during 7 consecutive days.
Step count | Change from baseline (T1) at 1 week after intervention (T2)
  Step count will be measured with an ActiGraph accelerometer during 7 consecutive days.
Step count | During 10-week intervention program
  Step count will be measured with a FitBit charge 4 during the 10-week intervention program
Resting heart rate | Baseline (T1)
  Resting heart rate will be measured for 10 minutes using a heart rate belt around the chest.
Blood pressure | Baseline (T1)
  Systolic and diastolic blood pressure will be measured with a blood pressure monitor.
Blood pressure | 1 week after intervention
  Systolic and diastolic blood pressure will be measured with a blood pressure monitor.
Sociodemographic and health-related characteristics | Baseline (T0)
  A general questionnaire assessing sociodemographic and health-related characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Van Oosterwijck, Principal Investigator — Department of Rehabilitation Sciences, Faculty of Health Sciences, Ghent University, Belgium
Locations (1):
- Ghent University, Ghent, Belgium

REFERENCES:
- [Background] Belavy DL, Van Oosterwijck J, Clarkson M, Dhondt E, Mundell NL, Miller CT, Owen PJ. Pain sensitivity is reduced by exercise training: Evidence from a systematic review and meta-analysis. Neurosci Biobehav Rev. 2021 Jan;120:100-108. doi: 10.1016/j.neubiorev.2020.11.012. Epub 2020 Nov 27. PMID 33253748
- [Background] Bernstein MS, Morabia A, Sloutskis D. Definition and prevalence of sedentarism in an urban population. Am J Public Health. 1999 Jun;89(6):862-7. doi: 10.2105/ajph.89.6.862. PMID 10358676
- [Background] Dhondt E, Danneels L, Van Oosterwijck S, Palmans T, Rijckaert J, Van Oosterwijck J. The influence of physical activity on the nociceptive flexion reflex in healthy people. Eur J Pain. 2021 Apr;25(4):774-789. doi: 10.1002/ejp.1708. Epub 2020 Dec 27. PMID 33290578
- [Background] Hakansson S, Jones MD, Ristov M, Marcos L, Clark T, Ram A, Morey R, Franklin A, McCarthy C, Carli LD, Ward R, Keech A. Intensity-dependent effects of aerobic training on pressure pain threshold in overweight men: A randomized trial. Eur J Pain. 2018 Nov;22(10):1813-1823. doi: 10.1002/ejp.1277. Epub 2018 Jul 11. PMID 29956398
- [Background] Hermans L, Van Oosterwijck J, Goubert D, Goudman L, Crombez G, Calders P, Meeus M. Inventory of Personal Factors Influencing Conditioned Pain Modulation in Healthy People: A Systematic Literature Review. Pain Pract. 2016 Jul;16(6):758-69. doi: 10.1111/papr.12305. Epub 2015 May 26. PMID 26011523
- [Background] Van Oosterwijck S, Meeus M, van Der Wekken J, Dhondt E, Billens A, Van Oosterwijck J. Physical Activity Is Predictive of Conditioned Pain Modulation in Healthy Individuals: A Cross-Sectional Study. J Pain. 2024 Nov;25(11):104639. doi: 10.1016/j.jpain.2024.104639. Epub 2024 Jul 18. PMID 39029881
- [Derived] Billens A, Hamelink T, Meeus M, Van Oosterwijck J. The influence of a moderate versus high intensity training program on central pain processing: a pilot feasibility study. Pain Manag. 2026 Feb 6:1-15. doi: 10.1080/17581869.2026.2626256. Online ahead of print. PMID 41649235